CLINICAL TRIAL: NCT00101400
Title: A Phase II Multicenter Uncontrolled Trial of BAY43-9006 in Subjects With Metastatic Breast Cancer.
Brief Title: BAY43-9006 - Phase II in Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100555
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Results first posted 2009-06-23 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-11

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Sorafenib 400 mg administered twice daily (b.i.d.)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib 400 mg administered twice daily (b.i.d.)

SUMMARY:
The purpose of this study is to evaluate the anti-cancer activity and safety of BAY43-9006 (Sorafenib) in patients, who suffer from an advanced breast tumour, which has spread to other organs of body despite treatment that the patient has received so far.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Women with prior histologically documented diagnosis of breast cancer
* Subjects with metastatic disease who have already received and failed at least one chemotherapy regimen for metastatic disease and, if ER/PgR +ve, have failed on at least adjuvant hormonal therapy
* Subjects for whom trastuzumab treatment is not indicated, no longer effective or refused by the subjects
* Four weeks since the last cytotoxic chemotherapy or clear evidence of progression on hormonal therapy
* Subjects who have at least one measurable lesion by CT (Computed Tomography) scan or MRI (Magnetic Resonance Imaging) according to modified WHO Tumour Response Criteria
* Subjects who have an Eastern Co-operative Oncology Group (ECOG) performance status of 0, 1 or 2
* Adequate bone marrow, liver and renal function as assessed by the following laboratory evaluations:

  * Hemoglobin > 9.0 g/dl
  * Absolute neutrophil count (ANC) > 1,500/mm3
  * Platelet count = 100,000/µl
  * Total bilirubin =1.5 x the upper limit of normal.
  * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) = 2.5 x upper limit of normal (=5 x upper limit of normal for subjects with liver involvement of their cancer)
  * Amylase and lipase = 1.5 x the upper limit of normal
  * Serum creatinine = 3.0 x the upper limit of normal
  * Prothrombin Time (PT) or International Normalized Ratio (INR) and Partial Thromboplastin Time (PTT) < 1.5 x upper limit of normal (subjects who receive anti-coagulation treatment with an agent such as warfarin or heparin will be allowed to participate provided that no evidence of underlying abnormality in these parameters exists)
* Subjects who give written informed consent prior to any study specific screening procedures with the understanding that the subject has the right to withdraw from the study at any time, without prejudice
* Life expectancy of at least 12 weeks
* Signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

* Previous malignancy (except for cervical carcinoma in situ, adequately treated basal cell carcinoma, or superficial bladder tumours [Ta, Tis and T1] or other malignancies curatively treated > 2 years prior to entry)
* Congestive heart failure > New York Heart Association (NYHA) Class II
* Cardiac arrhythmia requiring anti-arrhythmic (excluding beta blockers or digoxin)
* Active coronary artery disease or ischaemia
* Active clinically serious bacterial or fungal infections (> grade 2 National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 3)
* Known History of Human Immunodeficiency Virus (HIV) infection or chronic hepatitis B or C
* Metastatic brain or meningeal tumors unless the subject is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry. Also the patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable provided that the dose is stable for 1 month prior to and following screening radiographic study)
* Subjects with seizure disorders requiring medication (such as steroid or anti-epileptics)
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent
* Any condition that is unstable or which could jeopardize the safety of the subject and his/her compliance in the study. Pregnant or breast-feeding subjects. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug. Women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.

Excluded therapies include:

* Anti-cancer chemotherapy, hormonal therapy or immunotherapy during the study or within 4 weeks of study entry. Mytomicin or nitroureas should not be given within 6 weeks of study entry
* Significant surgery within 4 weeks prior to the start of study drug
* Any bone marrow transplant or stem cell rescue within 4 months of the start of study drug
* Radiotherapy during the study or within 3 weeks of the start of drug
* Use of biologic response modifiers, such as Granulocyte-Colony Stimulating Factor (G-CSF), within 3 weeks of study entry
* Investigational drug therapy outside of this trial during or within 30 days prior to start of the study drug
* Concomitant treatment with ketoconazole, itraconazole, ritonavir, or use of grapefruit juice
* Prior use of Raf-Kinase Inhibitors (RKI), Methyl Ethyl Ketone (MEK) or farnesyl transferase inhibitors
* Concomitant treatment or use of St. John's Wort
* Prior use of bevacizumab and all other drugs that target Vascular Endothelial Growth Factor (VEGF)/VEGF receptors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-02; Primary Completion 2006-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Germany (3):
  - Stuttgart, Baden-Wurttemberg
  - München, Bavaria
  - Frankfurt am Main, Hesse
- Italy (3):
  - Bologna
  - Milan
  - Parma

REFERENCES:
- [Result] Bianchi G, Loibl S, Zamagni C, Salvagni S, Raab G, Siena S, Laferriere N, Pena C, Lathia C, Bergamini L, Gianni L. Phase II multicenter, uncontrolled trial of sorafenib in patients with metastatic breast cancer. Anticancer Drugs. 2009 Aug;20(7):616-24. PMID 19739318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 03 Feb 2004 to 29 Jul 2004 by 3 centers in Germany and 4 centers in Italy.
Pre-assignment Details: 2 subjects were excluded during screening phase: 1 withdrawal of consent and 1 protocol violation.
Period: Treatment
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Started | 54 (Treated until disease progression, unacceptable sorafenib-related toxicity or withdrawal of consent.)
Completed | 54 (Reasons for treatment termination: 4 Adverse Events, 3 Deaths, 46 Progression, 1 Withdrawal.)
Not Completed | 0
Period: Survival Follow-Up
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Started | 51 (3 subjects died during previous period (completion as defined in protocol))
Completed | 44 (44 subjects reached endpoint (death); 7 subjects were still alive)
Not Completed | 7
Not completed — Alive | 7

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 0
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — 5-point, ordinal scale specifying patient's ability to perform activities from 0 (fully active) to 4 (completely disabled, no self-care)
  participants
    Grade 0: fully active | 30
    Grade 1: Restricted strenous activity, ambulatory | 22
    Grade 2: Ambulatory, difficulty in walking | 2
    Grade 3: Limited self-care, partly confined to bed | 0
    Grade 4: Completely disabled, no self-care | 0
Stage of disease at study entry (Tumor, Nodules, Metastasis (TNM) classification) [Number; unit: participants] — Categorized information on tumor size, lymph node involvement and metastases. Overall cancer staging (I - IV) is based on the TNM categories. The higher the overall stage, the more advanced the cancer is.
  participants
    Stage I | 0
    Stage II | 0
    Stage III | 0
    Stage IV -most advanced | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Response (Complete or Partial)
Description: Number of subjects with metastatic breast cancer treated with single agent BAY43-9006 who had best overall response assessed as complete response (CR) or partial response (PR) as per Modified World Health Organization (WHO) Tumor Response Criteria.
Time Frame: Until 30 days after termination of active therapy
Population: Intent to treat population consisted of subjects who received at least 1 dose of sorafenib.
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 54
participants
  Complete response (CR) | 0
  Partial response (PR) | 1
  Stable disease (SD) | 20
  Progressive disease (PD) | 31
  Not evaluated | 2

2. Secondary Outcome: Time to Progression
Description: Time from start of treatment until progression was first documented.
Time Frame: Until progression occurs
Population: Of the intent to treat population, 4 subjects died before assessment of progression; for 1 subject the progression date not available; and 1 subject was lost to follow-up.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 48
days | 58 [52 to 112]

3. Secondary Outcome: Time to Objective Response
Description: Defined only for subjects achieving objective tumor response from start of treatment to the date when confirmed PR or CR was first documented according to the Modified WHO Tumor Response Criteria.
Time Frame: Until objective response occurs
Population: 1 subject out of 54 achieved PR.
Measure: Number; unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 1
days | 145

4. Secondary Outcome: Overall Response Duration
Description: Overall response duration was defined only for subjects achieving confirmed objective response (PR or CR). It was measured from start of treatment to the date when progressive disease was first objectively documented.
Time Frame: Time from PR or CR to progression
Population: 1 subject out of 54 achieved PR.
Measure: Number; unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 1
days | 256

5. Secondary Outcome: Survival Time
Description: After the end of treatment visit (30 days after the last dose), the subjects were monitored every 3 months for survival (visits/phone calls).
Time Frame: Start of treatment to death
Population: Intent to treat population consisting of subjects who received at least 1 dose of sorafenib.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 54
days | 259 [177 to 323]

6. Secondary Outcome: Number of Subjects With Stable Disease up to Cycle 4
Description: Number of subjects who had not responded to treatment but had stable disease up to cycle 4.
Time Frame: Until 30 days after termination of active therapy
Population: Intent to treat population consisting of subjects who received at least 1 dose of sorafenib.
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 54
participants | 12

ADVERSE EVENTS:
Description: Acronyms used: Gastrointestinal (GI), Common Terminology Criteria for Adverse Events (CTCAE), Not Otherwise Specified (NOS), Central nervous system (CNS), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Gammaglutamyltransferase (GGT).
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Serious Adverse Events (participants affected / at risk) | 22/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=54)
Hemoglobin (Blood and lymphatic system disorders) | 1
Coagulation - Other (Blood and lymphatic system disorders) | 1
Supraventricular Arrhythmia, Supraventricular Tachycardia (Cardiac disorders) | 1
Cardiac General - Other (Cardiac disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Perforation, GI, Colon (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death Not Associated With CTCAE Term, Disease Progression NOS (General disorders) | 3
Fever (General disorders) | 1
Fatigue (General disorders) | 7
Pain, Back (General disorders) | 2
Pain, Chest/Thorax NOS (General disorders) | 1
Pain, Abdomen NOS (General disorders) | 3
Pain, Head/Headache (General disorders) | 1
Liver Dysfunction (Hepatobiliary disorders) | 3
Hepatobiliary - Other (Hepatobiliary disorders) | 2
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 3
Neuropathy: Motor (Nervous system disorders) | 1
CNS Necrosis (Nervous system disorders) | 1
Neurology - Other (Nervous system disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Shortness Of Breath) (Respiratory, thoracic and mediastinal disorders) | 7
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=54)
Neutrophils (Blood and lymphatic system disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 5
Platelets (Blood and lymphatic system disorders) | 5
Leukocytes (Blood and lymphatic system disorders) | 3
Dermal Change (Blood and lymphatic system disorders) | 3
Edema: Limb (Blood and lymphatic system disorders) | 7
Hypertension (Cardiac disorders) | 3
Cardiac General - Other (Cardiac disorders) | 3
Anorexia (Gastrointestinal disorders) | 29
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 14
Dysphagia (Gastrointestinal disorders) | 7
Gastritis (Gastrointestinal disorders) | 9
Mucositis (Clinical Exam), Oral Cavity (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 11
Fever (General disorders) | 7
Insomnia (General disorders) | 6
Fatigue (General disorders) | 27
Weight Loss (General disorders) | 3
Constitutional Symptoms - Other (General disorders) | 5
Pain, Back (General disorders) | 4
Pain, Extremity - Limb (General disorders) | 4
Pain, Abdomen NOS (General disorders) | 9
Pain, Head/Headache (General disorders) | 6
Pain, Joint (General disorders) | 4
Pain, Bone (General disorders) | 9
Pain, Other (General disorders) | 16
Pain, Liver (General disorders) | 3
Pain, Stomach (General disorders) | 6
Hepatobiliary - Other (Hepatobiliary disorders) | 3
Infection - Other (Infections and infestations) | 6
Alkaline Phosphatase (Metabolism and nutrition disorders) | 7
ALT (Metabolism and nutrition disorders) | 10
AST (Metabolism and nutrition disorders) | 8
GGT (Metabolism and nutrition disorders) | 7
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 5
Mood Alteration, Anxiety (Nervous system disorders) | 4
Confusion (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 6
Neurology - Other (Nervous system disorders) | 5
Neuropathy: Sensory (Nervous system disorders) | 7
Somnolence (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Shortness Of Breath) (Respiratory, thoracic and mediastinal disorders) | 14
Alopecia (Skin and subcutaneous tissue disorders) | 9
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 13
Nail Changes (Skin and subcutaneous tissue disorders) | 3
Dermatology - Other (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 15
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 21
Flushing (Skin and subcutaneous tissue disorders) | 4
Hemorrhage Pulmonary, Nose (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
Subjects had advanced disease and were heavily pretreated. Not all adverse events mentioned were assessed as drug-related. NCI-CTCAE was translated to Medical Dictionary for Regulatory Activities (MedDRA) for System Organ Classes (SOCs) only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days